CLINICAL TRIAL: NCT00902538
Title: Add-on Study of Hydrochlorothiazide in Patients With Moderate to Severe Hypertension Not Achieving Target Blood Pressure on Olmesartan/Amlodipine Alone
Brief Title: Hydrochlorothiazide as add-on to Olmesartan/Amlodipine in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS8635-A-E303
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2012-02

CONDITIONS: Essential Hypertension
Keywords: Add on treatment; essential hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Amlodipine; olmesartan; Hydrochlorothiazide; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Olmesartan (OLM) 40mg-Amlodipine (AML) 10mg (Experimental): The participants in this arm received these 2 drugs for the 8-week, single-blind, run-in Period 1. Participants could then randomized to this same combination for an additional 8 weeks in the double-blind, Period 2.
  Interventions: Drug: Olmesartan medoxomil 40 mg - Amlodipine 10 mg
- Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 12.5mg (Experimental): Participants could start receiving this combination in randomized, double-blind, 8-week Period 2. This combination was continued into single-blind, 8-week Period 3 for all participants entering Period 3.
  Interventions: Drug: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 12.5mg
- Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 25mg (Experimental): Participants could start receiving this combination in randomized, double-blind, 8- week Period 2.
  Interventions: Drug: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 25mg
- OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg (Responders) (Experimental): Participants who meet their blood pressure goals in Period 3 and continued into the 8-week, double-blind Period 4 continued to receive this combination.
  Interventions: Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg
- OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg (Non-responders) (Experimental): Participants finishing Period 3, but, who did not meet their blood pressure goals could receive this combination in the double-blind, randomized, Period 4
  Interventions: Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg
- OLM 40mg-AML 10mg-Hydrochlorothiazide 25mg (Non-responders) (Experimental): Participants finishing Period 3, but, who did not meet their blood pressure goals could receive this combination in the double-blind, randomized, Period 4
  Interventions: Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 25mg

INTERVENTIONS:
Drug: Olmesartan medoxomil 40 mg - Amlodipine 10 mg — Oral tablets containing Olmesartan medoxomil-Amlodipine 40-10 mg, given once daily
  Arms: Olmesartan (OLM) 40mg-Amlodipine (AML) 10mg
Drug: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 12.5mg — Coated, oral tablets containing Olmesartan 40mg-Amlodipine 10mg + 1 Hydrochlorothiazide 12.5mg oral tablet + 1 Hydrochlorothiazide 12.5mg oral, placebo tablet. All tablets are given once a day.
  Arms: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 12.5mg
Drug: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 25mg — Coated, oral tablets containing Olmesartan 40mg-Amlodipine 10mg + 2 Hydrochlorothiazide 12.5mg oral tablets. All tablets are given once a day.
  Other Names: Olmesartan 40mg-Amlodipine 10mg tablet + 2 Hydrochlorothiazide 12.5mg tablets
  Arms: Olmesartan 40mg-Amlodipine 10mg-Hydrochlorothiazide 25mg
Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg — Coated, oral tablets containing Olmesartan 40mg-Amlodipine 10mg + 1 Hydrochlorothiazide 12.5mg oral tablet + 1 Hydrochlorothiazide 12.5mg oral, placebo tablet. All tablets are given once a day.
  Arms: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg (Responders)
Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg — Coated, oral tablets containing Olmesartan 40mg-Amlodipine 10mg + 1 Hydrochlorothiazide 12.5mg oral tablet + 1 Hydrochlorothiazide 12.5mg oral, placebo tablet. All tablets are given once a day.
  Arms: OLM 40mg-AML 10mg-Hydrochlorothiazide 12.5mg (Non-responders)
Drug: OLM 40mg-AML 10mg-Hydrochlorothiazide 25mg — Coated, oral tablets containing Olmesartan 40mg-Amlodipine 10mg + 2 Hydrochlorothiazide 12.5mg oral tablet. All tablets are given once a day.
  Arms: OLM 40mg-AML 10mg-Hydrochlorothiazide 25mg (Non-responders)

SUMMARY:
Both Olmesartan (OLM)/Amlodipine (AML) combination and Hydrochlorothiazide (HCTZ) have proven to be efficacious and safe in lowering blood pressure, but may not always be sufficient. This study is to test efficacy and safety of the combination of OLM/AML and HCTZ in hypertensive patients whose blood pressure is not adequately controlled with OLM/AML alone. The following treatments will be included in the trial: OLM 40mg/AML 10mg; OLM 40mg/AML 10 mg/HCTZ 12.5 mg; OLM 40 mg/AML 10 mg/HCTZ 25 mg. The trial has four periods. The treatments that will be used are as follows:

Period 1 - OLM 40mg/AML 10mg; Period 2 - OLM 40mg/AML 10mg or OLM 40mg/AML 10 mg/HCTZ 12.5 mg or OLM 40 mg/AML 10 mg/HCTZ 25 mg; Period 3 - OLM 40mg/AML 10 mg/HCTZ 12.5 mg; Period 4 - Period 3 responders: OLM 40mg/AML 10 mg/HCTZ 12.5 mg; Period 4 - Period 3 non-responders: OLM 40mg/AML 10 mg/HCTZ 12.5 mg or OLM 40 mg/AML 10 mg/HCTZ 25 mg

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older.
* Mean trough seated systolic blood pressure (SeSBP) of ≥ 160/100 mmHg (SeSBP of ≥ 160 mmHg and seated diastolic blood pressure (SeDBP) ≥ 100 mmHg) at screening if not currently on antihypertensive medication (e.g. newly diagnosed subjects)

OR:

For subjects on monotherapy: mean trough SeSBP of ≥ 150/95 mmHg (SeSBP of ≥ 150 mmHg and SeDBP ≥ 95 mmHg) at screening

OR:

For subjects on any combination of antihypertensive medications that includes either hydrochlorothiazide or amlodipine or olmesartan for a duration of at least four weeks: mean trough SeSBP of ≥ 140/90 mmHg (SeSBP of ≥ 140 mmHg and SeDBP ≥ 90 mmHg) at screening

OR:

For subjects on any other combination of antihypertensive medications that includes neither hydrochlorothiazide, amlodipine nor olmesartan: mean trough SeSBP ≥ 160 mmHg, mean trough SeDBP ≥ 100mmHg, at the end of the taper-off period

* Subject freely signs the Informed Consent Form (ICF) after the nature of the study and the disclosure of his/her data has been explained.
* Female subjects of childbearing potential must be using adequate contraception (female of childbearing potential is defined as one who has not been postmenopausal for at least one year, or has not been surgically sterilised, or has not had a hysterectomy at least three months prior to the start of this study [Visit 1]). Females taking oral contraceptives should have been on therapy for at least three months. Adequate contraceptives include hormonal intra-uterine devices, hormonal contraceptives (oral, depot, patch or injectable), and double barrier methods such as condoms or diaphragms with spermicidal gel or foam. If a female becomes pregnant during the study, she has to be withdrawn immediately.

Exclusion Criteria:

* Female subjects of childbearing potential who are pregnant or lactating.
* Subjects with serious disorders which may limit the ability to evaluate the efficacy or safety of the investigational products, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematological or oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic subjects.
* Subjects having a history of the following within the last six months: myocardial infarction (MI), unstable angina pectoris, percutaneous coronary intervention, heart failure, hypertensive encephalopathy, cerebrovascular accident (stroke), or transient ischaemic attack.
* Subjects with clinically significant abnormal laboratory values at Screening, including subjects with one or more of the following:

  * Aspartate aminotransferase (AST) > 3 times upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) > 3 times ULN
  * Gamma-glutamyltransferase (GGT) > 3 times ULN
  * Potassium above ULN (unless high value is due to haemolytic blood sample)
* Subjects with secondary hypertension of any aetiology such as renal disease, phaeochromocytoma, or Cushing's syndrome.
* Subjects with contraindication to olmesartan, amlodipine, hydrochlorothiazide, or any of the excipients.
* Subjects with a mean SeSBP > 200 mmHg or mean SeDBP > 115 mmHg or bradycardia (heart rate < 50 beats/min at rest documented by mean radial pulse rate [PR] or electrocardiogram [ECG]) at Screening (Visit 1) or immediately before taking Period I study medication (Visit 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2204 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (117):
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- Belgium (6):
  - Antwerp
  - Lauwe
  - Leuven
  - Liège
  - Massemen
  - Oostham
- Bulgaria (5):
  - Haskovo
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Czechia (9):
  - Bílovec
  - Brno
  - Havlíčkův Brod
  - Hodonín
  - Kladno
  - Kolín
  - Ostrava
  - Ostrava-Vitkovice
  - Prague
- Denmark (4):
  - Copenhagen
  - Frederiksberg
  - Næstved
  - Roskilde
- France (15):
  - Albi
  - Angers
  - Brest
  - Cambrai
  - Créteil
  - Dijon
  - Dinard
  - Lyon
  - Nancy
  - Pessac
  - Roubaix
  - Strasbourg
  - Tiercé
  - Vandœuvre-lès-Nancy
  - Villefranche-de-Rouergue
- Germany (9):
  - Berlin
  - Dresden
  - Einbeck
  - Hamburg
  - Magdeburg
  - München
  - Straßkirchen
  - Villingen-Schwenningen
  - Wermsdorf
- Netherlands (6):
  - Almere Stad
  - Beek en Donk
  - Doetinchem
  - Groningen
  - Losser
  - Maastricht
- Poland (11):
  - Bytom
  - Gdansk
  - Katowice
  - Krakow
  - Piotrkow Trybunalski
  - Puławy
  - Siemianowice Śląskie
  - Tarnów
  - Torun
  - Warsaw
  - Wroclaw
- Romania (9):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Oradea
  - Piteşti
  - Târgovişte
  - Târgu Mureş
  - Timișoara
- Russia (10):
  - Moscow
  - Novosibirsk
  - Orenburg
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tomsk
  - Yaroslavl
  - Yekaterinburg
- Slovakia (6):
  - Banska Bysterica
  - Brastislava
  - Dolný Kubín
  - Košice
  - Prešov
  - Šahy
- Spain (12):
  - La Gineta, Albacete
  - La Roda, Albacete
  - Port de Sagunt, Valencia
  - Alicante
  - Barcelona
  - Elche
  - Granada
  - Madrid
  - Palma de Mallorca
  - Seville
  - Valencia
  - Vizcaya
- Ukraine (12):
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Lviv
  - Mykolayiv
  - Odesa
  - Simferopol
  - Uzhhorod
  - Vinnytsia
  - Yalta

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant visit was 29 April 2009. The last participant follow up was 07 September 2010
Pre-assignment Details: The number of subjects entering Period 2 was only 808 because 1278 did not meet the entry criteria.
Groups:
- Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg: The participants in this arm received Olmesartan(OLM) 40 mg-Amlodipine(AML) 10 mg oral tablets, once a day, for the 8-week, single-blind, run-in Period 1. Then in Period 2, participants would be randomized to this same combination or have hydrochlorothiazide oral tablets (12.5 or 25 mg) added for an additional 8 weeks. All medication is given once a day.
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5: Participants could start receiving OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 oral tablets given once daily in randomized, double-blind, 8-week Period 2. This combination was continued into single-blind, 8-week Period 3 for all participants entering Period 3.
- OLM 40-AML 10-HCTZ 25: Participants could start receiving OLM 40-AML 10-HCTZ 25 oral tablets, given once daily, in randomized, double-blind, 8- week Period 2.
- OLM 40-AML 10-HCTZ 12.5 (Responders): Participants who meet their blood pressure goals (responded) in Period 3 and continued into 8-week, double-blind Period 4 continued to receive OLM 40-AML 10-HCTZ 12.5 oral tablets given once daily.
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders): Participants finishing Period 3, but, who did not meet their blood pressure goals (non-responders) could receive OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 oral tablets, given once daily, in double-blind, randomized, Period 4.
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders): Participants finishing Period 3, but, who did not meet their blood pressure goals (non-responders) could receive OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 oral tablets, given once daily, in double-blind, randomized, Period 4
Period: 1-Single-blind, Run-in, Single-Treatment
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25 | OLM 40-AML 10-HCTZ 12.5 (Responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Started | 2204 | 0 | 0 | 0 | 0 | 0
Completed | 2086 | 0 | 0 | 0 | 0 | 0
Not Completed | 118 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 49 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 30 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 22 | 0 | 0 | 0 | 0 | 0
Not completed — Other Reason | 13 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0 | 0
Period: 2-Randomized Double-blind 3 Treatments
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25 | OLM 40-AML 10-HCTZ 12.5 (Responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Started | 269 (Only 808 began Period 2 because the others finishing Period 1 did not meet the entry criteria.) | 269 | 270 | 0 | 0 | 0
Completed | 260 | 263 | 262 | 0 | 0 | 0
Not Completed | 9 | 6 | 8 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0 | 0 | 0
Period: 3-Single-blind, Single Treatment
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25 | OLM 40-AML 10-HCTZ 12.5 (Responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Started | 0 | 782 (Number starting is < total completing previous arm since 3 subjects did not receive at least 1 dose.) | 0 | 0 | 0 | 0
Completed | 0 | 767 | 0 | 0 | 0 | 0
Not Completed | 0 | 15 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Period: 4-Randomized Double-blind 2 Treatments
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25 | OLM 40-AML 10-HCTZ 12.5 (Responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Started | 0 | 0 | 0 | 467 (Period 3 responders were continued on OLM 40-AML 10-HCTZ 12.5) | 97 (Period 3 non-responders were randomized to OLM 40-AML 10-HCTZ 12.5 or 25 in a 2:1 ratio) | 197
Completed | 0 | 0 | 0 | 458 | 95 | 196
Not Completed | 0 | 0 | 0 | 9 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg: The participants in this arm received these 2 drugs for the 8-week, single-blind, run-in Period 1. Participants could then randomized to this same combination for an additional 8 weeks in the double-blind, Period 2.
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5: Participants could start receiving this combination in randomized, double-blind, 8- week Period 2. This combination was continued into single-blind, 8-week Period 3 for all participants entering Period 3
- OLM 40-AML 10-HCTZ 25: Participants could start receiving this combination in randomized, double-blind, 8- week Period 2.
- Total: Total of all reporting groups
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25 | Total
Number analyzed (Participants) | 269 | 269 | 270 | 808
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.56) | 56.5 (10.25) | 54.9 (10.44) | 55.8 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 104 | 116 | 339
  Male | 150 | 165 | 154 | 469
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 269 | 269 | 269 | 807
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 87.8 (18.14) | 88.2 (16.03) | 88.5 (16.28) | 88.2 (16.83)
Height [Mean (Standard Deviation); unit: cm] | 169.9 (9.74) | 170.5 (9.11) | 170.4 (8.98) | 170.3 (9.27)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.27 (4.90) | 30.30 (4.65) | 30.44 (4.87) | 30.34 (4.80)
Obesity [Number; unit: Participants] — Number of participants whose Body Mass Index (BMI) is <30 kg/m^2 or whose number is >=30 kg/m^2. Only 806 participants had their BMI measured.
  Participants
    Body Mass Index < 30 kg/m^2 | 138 | 142 | 133 | 413
    Body Mass Index >= 30 kg/m^2 | 131 | 125 | 137 | 393

OUTCOME MEASURES:

1. Primary Outcome: Change in Seated Diastolic Blood Pressure (SeDBP) of the Triple Combinations OM/AML/HCTZ 40/10/12.5 and 40/10/25 mg vs. OM/AML 40/10 mg
Description: Three cuff blood pressure measurements were taken at each visit.
Time Frame: baseline (8 weeks) to 16 weeks
Population: The Full Analysis Set 1 included 806 randomized subjects who received at least 1 dose of double-blind study medication in Period II and provided at least 1 SeDBP measurement in Period II: 269 subjects in the OM/AML 40/10 mg group, 268 subjects in the OM/AML/HCTZ 40/10/12.5 mg group, and 269 subjects in the OM/AML/HCTZ 40/10/25 mg group.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5: Participants could start receiving this combination in randomized, double-blind, 8-week Period 2. This combination was continued into single-blind, 8-week Period 3 for all participants entering Period 3.
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 269 | 268 | 269
mm Hg | -6.1 (0.55) | -7.1 (0.55) | -8.9 (0.55)
Statistical Analysis 1: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5; Test type: Superiority or Other; p = 0.1187, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Change in Seated Systolic Blood Pressure (SeSBP) of the Triple Combinations OM/AML/HCTZ 40/10/12.5 and 40/10/25 mg vs. OM/AML 40/10 mg
Description: Three cuff blood pressure measurements were taken at each visit.
Time Frame: baseline (8 weeks) to week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 269 | 268 | 269
mm Hg | -6.9 (0.76) | -8.6 (0.77) | -10.5 (0.77)
Statistical Analysis 1: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5; Test type: Superiority or Other; p = 0.0425, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p < 0.0001, ANCOVA

3. Secondary Outcome: Number of Subjects Achieving Blood Pressure (BP) Goal at Week 16.
Description: Achieving blood pressure goal is defined as seated blood pressure <140/90 mm Hg; 130/80 mm Hg for participants with diabetes and/or other chronic renal and/or chronic cardiovascular disease. Three cuff blood pressure measurements were taken at each visit.
Time Frame: baseline (week 8) to week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 269 | 268 | 269
Participants | 65 | 79 | 111
Statistical Analysis 1: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5; Test type: Superiority or Other; p = 0.1939, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in 24-hour Diastolic Blood Pressure (DBP) Assessed by 24-hour Ambulatory Blood Pressure Measurement (ABPM).
Description: Three cuff blood pressure measurements were taken at each visit.
Time Frame: Baseline (8 weeks) to 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 269 | 268 | 269
mm Hg | -2.1 (0.52) | -4.0 (0.52) | -5.3 (0.52)
Statistical Analysis 1: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5; Test type: Superiority or Other; p = 0.0009, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p < 0.0001, ANCOVA

5. Secondary Outcome: Change in 24-hour Systolic Blood Pressure Assessed by 24-hour Ambulatory Blood Pressure Measurement.
Description: Three cuff blood pressure measurements were taken at each visit.
Time Frame: Baseline (8 weeks) to 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 269 | 268 | 269
mm Hg | -1.9 (0.75) | -5.1 (0.75) | -6.6 (0.75)
Statistical Analysis 1: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p < 0.0001, ANCOVA

6. Secondary Outcome: In Non-responders, the Change in Seated Diastolic Blood Pressure Associated With the Triple Combinations OM/AML/HCTZ 40/10/12.5 and 40/10/25 mg.
Description: Change in seated diastolic blood pressure from the beginning to the end of Period 4. Three cuff blood pressure measurements were taken at each visit.
Time Frame: week 24 to week 32
Population: The analysis population includes those participants who had blood pressure values at both the beginning and end of Period 4.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders); OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders): Participants finishing Period 3, but, who did not meet their blood pressure goals could receive this combination in the double-blind, randomized, Period 4
Arm/Group | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Number analyzed (Participants) | 96 | 196
mm Hg | -6.7 (0.84) | -7.9 (0.69)
Statistical Analysis 1: Comparison: OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders); Test type: Superiority or Other; p = 0.1611, ANCOVA

7. Secondary Outcome: In Non-responders, the Change in Seated Systolic Blood Pressure Associated With the Triple Combinations OM/AML/HCTZ 40/10/12.5 and 40/10/25 mg.
Description: Change in seated systolic blood pressure from the beginning to the end of Period 4. Three cuff blood pressure measurements were taken at each visit.
Time Frame: week 24 to week 32
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Number analyzed (Participants) | 96 | 196
mm Hg | -5.5 (1.10) | -7.8 (0.89)
Statistical Analysis 1: Comparison: OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders); Test type: Superiority or Other; p = 0.0451, ANCOVA

8. Secondary Outcome: In Non-responders, the Number of Subject Meeting Their Blood Pressure Goals Associated With the Triple Combinations OM/AML/HCTZ 40/10/12.5 and 40/10/25 mg.
Description: The number of non-responding participants who achieved their blood pressure goals at the end of Period 4. Achieving blood pressure goal is defined as seated blood pressure <140/90 mm Hg; 130/80 mm Hg for participants with diabetes and/or other chronic renal and/or chronic cardiovascular disease. Three cuff blood pressure measurements were taken at each visit.
Time Frame: week 24 to week 32
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders)
Number analyzed (Participants) | 96 | 196
Participants | 31 | 89
Statistical Analysis 1: Comparison: OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (Non-responders) vs OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 25 (Non-responders); Test type: Superiority or Other; p = 0.0412, ANCOVA

9. Secondary Outcome: In Non-responders, the Change in 24-hour Diastolic Blood Pressure Assessed by 24-hour Ambulatory Blood Pressure Measurement.
Description: In non-responders, the change in 24-hour diastolic blood pressure assessed by 24-hour ambulatory blood pressure measurement from the beginning to the end of Period 4.
Time Frame: Week 16 to week 32
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 96 | 196
mm Hg | -2.2 (0.96) | -4.4 (0.81)
Statistical Analysis 1: Comparison: OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p = 0.0253, ANCOVA

10. Secondary Outcome: In Non-responders, the Change in 24-hour Systolic Blood Pressure Assessed by 24-hour Ambulatory Blood Pressure Measurement.
Description: In non-responders, the change in 24-hour systolic blood pressure assessed by 24-hour ambulatory blood pressure measurement from the beginning to the end of Period 4.
Time Frame: Week 16 to week 32
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Number analyzed (Participants) | 96 | 196
mm Hg | -0.4 (1.44) | -4.3 (1.21)
Statistical Analysis 1: Comparison: OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 vs OLM 40-AML 10-HCTZ 25; Test type: Superiority or Other; p = 0.0063, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening to 14 days after the last dose of study medication. Adverse events are reported for week 1 through week 16.
Arm/Group | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 | OLM 40-AML 10-HCTZ 25
Serious Adverse Events (participants affected / at risk) | 18/2204 | 15/269 | 3/270
Other Adverse Events (participants affected / at risk) | 113/2204 | 7/269 | 7/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg (N=2204) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (N=269) | OLM 40-AML 10-HCTZ 25 (N=270)
Ankle fracture (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flbrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral aterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pseudoathrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophelibitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olmesartan(OLM) 40 Mg-Amlodipine(AML) 10 mg (N=2204) | OLM 40-AML 10-Hydrochlorothiazide (HCTZ) 12.5 (N=269) | OLM 40-AML 10-HCTZ 25 (N=270)
Oedema peripheral (General disorders) | 113 (113) | 7 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A site may not publish results until after a multi-center publication has been submitted for publication or until one year after the study has ended, whichever occurs first. Then, the site will have the opportunity to publish the results, provided that Daiichi Sankyo Europe has had the opportunity to review and comment on the site's proposed publication prior to its being submitted for publication with the advice of company patent council and in accord with needs for subject protection.